CLINICAL TRIAL: NCT06842056
Title: Multicentric Multinational Observational Study to Describe the Shift in Stage at Diagnosis of Lung Cancer. No Direct Recruitment of Patients or Administration of Study Medication.
Brief Title: Multinational Observational Study to Describe Diagnostic Stage Shift in Patients With Lung Cancer Using Medical Records
Acronym: DIASTAG
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133HR00049
Record Dates: First submitted 2025-02-07; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Aggregate data; Non small cell lung cancer; data extraction; Early stage; Locally advanced; Late stage
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multinational observational study to describe diagnostic stage shift in patients with lung cancer using medical records. Increased lung cancer screening programs and increased utilization of other screening modalities such as large increase in community chest radiography referral rates in response to public awareness campaigns, as well as unintentional detections through cardiac CT(computed tomography) angiograms, or screening for coronary disease may help in detecting the disease at earlier curable stages. Availability and increased access to novel therapies increase the likelihood of an early-stage diagnosis aiming for improved survival.

DETAILED DESCRIPTION:
This is a multicentric, multinational, observational study to describe the shift in stage at diagnosis of lung cancer over the time- period from baseline year to EOS (end of study). The study will be implemented in the AstraZeneca International Region (ie, non-US, non-European countries). The participating countries and sites will be selected based on the availability and accessibility of secondary data sources such as lung cancer databases or EMR (electronic medical records) in the target countries. Once countries and databases are selected, the protocol will be adapted for the specific country including details about the patient databases. The study will be conducted in compliance with the local legal, ethical, and regulatory requirements of the selected countries. The study-specific data will be extracted from the databases and recorded using eCRF (electronic case report form). This study does not involve direct recruitment of the patients. Aggregated data from the databases for each consecutive year starting from the baseline year until EOS, of patients with lung cancer meeting the inclusion criteria will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult female and male patients ≥18 years old.
* Confirmed diagnosis of lung cancer (either cytologically or histologically)

Exclusion Criteria:

* Patients presenting with recurrent or relapsed lung cancer.
* Patients with a concomitant cancer at the time of diagnosis of lung cancer, except for nonmetastatic nonmelanoma skin cancers, or in situ or benign neoplasms: a cancer will be considered concomitant if it occurs within 5 years of lung cancer diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study does not involve direct recruitment of the patients. Aggregated data from the databases for each consecutive year starting from the baseline year until End of study. Patients with lung cancer meeting the following criteria will be included in the study.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Early stage (stage I and II with [N0]) | 5 years
  Number and percentage of patients diagnosed with Early stage (stage I and II with [N0]) from baseline year until EOS
Locally advanced (stage II and III [N+]) | 5 years
  Number and percentage of patients diagnosed with Locally advanced (stage II and III [N+]) from baseline year until EOS
Late stage (stage IV [M1]) | 5 years
  Number and percentage of patients diagnosed with Late stage (stage IV [M1]) from baseline year until EOS

SECONDARY OUTCOMES:
screening based on clinical presentation | 5 years
  Number and percentage of patients with modalities of diagnosis and screening at the yearly data cut-off based on clinical presentation
Incidental diagnosis | 5 years
  Number and percentage of patients with Incidental diagnosis o Through screening program (Yes/No) If yes, screening modality (LDCT/ sputum microscopy/ chest X-ray/ any other)
TNM staging | 5 years
  Number and percentage of patients presenting with TNM staging according to AJCC 8th edition (Aberle, 2011;Kutob, 2019) or staging by alternative lung cancer staging system
Histological type | 5 years
  Number and percentage of patients presenting with lung cancer diagnosis. Histological type

OTHER OUTCOMES:
Age categories | 5 years
  Relationship between the diagnosis at early stage and following characteristics - Age categories
smoking categories. | 5 years
  Relationship between the diagnosis at early stage with smoking categories

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/